CLINICAL TRIAL: NCT02463448
Title: Autologous Muscle Derived Cells for Underactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jason Gilleran (Other)
Responsible Party: Sponsor-Investigator, Jason Gilleran, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-134
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Urinary Retention; Urinary Incontinence
Keywords: Underactive Bladder
MeSH Terms: conditions — Urinary Retention; Urinary Incontinence; Urinary Bladder, Underactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Muscle Derived Cells (Experimental): Autologous Muscle Derived Cells are obtained by needle biopsy from the subject's own thigh muscle. These cells are sent to a special lab for growth and processing. When ready the cells are sent to the treatment location for injection into the bladder wall.
  Interventions: Biological: Autologous Muscle Derived Cells

INTERVENTIONS:
Biological: Autologous Muscle Derived Cells — A small sample of the subject's own thigh muscle is obtained by needle biopsy. The biopsy sample is sent to Cook Myosite, Inc. for growth and processing. When the sample cell dosage is achieved the cells are frozen and sent back to the treatment site. The cells are thawed, diluted and injected under lighted instrumentation and visualization into about 30 sites in the bladder wall.

SUMMARY:
This is a prospective, open-label, Phase 1, single center study evaluating the safety and efficacy of Autologous Muscle Derived Cells as a treatment for chronic Underactive Bladder.

DETAILED DESCRIPTION:
Subject that meet inclusion and exclusion criteria will be consented and enrolled in this study. Initial screening includes blood and urine testing, questionnaires, physical examination, specialized bladder function testing and review of medical history. At the next visit a small sample of each subject's own thigh muscle is obtained by needle biopsy. This cell biopsy is sent to a specialized lab for growth and processing. Approximately ten weeks later the frozen cells will be sent back to the treatment site for thawing, diluting and injection under lighted instrumentation into the subject's bladder wall. The subject will be followed for 6 months and at that time may be eligible for a second injection of cells. The study doctor will determine if the second injection may be beneficial to the subject. All subjects will be followed for up to 12 months. The follow-up assessments at 12 months will include questionnaires, urine and blood testing, specialized bladder function testing and visualizing the inside of the bladder with a lighted instrument.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, at least 18 years of age
2. History of Underactive Bladder (UAB) for at least 6 months documented in the medical record
3. Recurring UAB symptoms
4. Subjects unresponsive to relief symptoms of UAB with previous use of medications and/or other treatments
5. Voiding difficulty (complains of difficulty emptying the bladder)
6. Post void residual greater than or equal to 150 mL
7. Total UAB Questionnaire Score greater than or equal to 3
8. Females of child-bearing potential agree to use a reliable form of birth control for the entire study duration
9. Willing and capable of understanding and complying with all requirements of the protocol, including proper completion of the voiding diaries and self-administered questionnaires

Exclusion Criteria:

1. Pregnant, plans to become pregnant or lactating
2. History of bleeding diathesis, uncorrectable coagulopathy, or would refuse a blood transfusion
3. Currently on anticoagulant therapy
4. Obvious neurological impairment
5. Known allergy or hypersensitivity to bovine proteins or allergens, gentamicin sulfate, ampicillin, and/or lidocaine that medically warrants exclusion as determined by the physician
6. Simultaneously participating in another investigational drug or device study or use of any investigational drug(s) or therapeutic device(s) within 3 months preceding enrollment
7. Has been treated with an investigational device, drug, or procedure for UAB within the last 6 months.
8. Medical condition or disorder that may limit life expectancy or that may cause protocol deviations (e.g. unable to perform self-evaluations and/or accurately report medical history, urinary symptoms, and/or data)
9. History of cancer in pelvic organs, ureters, or kidneys or any cancer that has undergone treatment within the past 12 months
10. Compromised immune system due to disease state, chronic corticosteroid use, or other immunosuppressive therapy
11. History of radiation therapy to the bladder
12. Tests positive for Hepatitis B (Hepatitis B Surface Antigen), and Anti-Hepatitis B Core Total Antibody, Hepatitis C (Anti-Hepatitis C virus enzyme immunoassay, Human Immunodeficiency Virus (HIV Type I and 2 Antibodies), and/or Syphilis
13. Abnormal renal function
14. An active urinary tract infection as evidenced by positive urine culture
15. Taking medication(s) that affect urination (e.g. medically necessary, stable drugs) such as prescription drugs, over-the-counter drugs, or dietary supplements, including herbal supplements and those taken with teas
16. Requires concomitant use of or treatment with immunosuppressive agents
17. Pelvic organ prolapse beyond the introitus (e.g., cystocele, rectocele)
18. Abnormal bladder capacity (i.e., less than 100 mL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gilleran, MD, Principal Investigator — Beaumont Health
Locations (1):
- Beaumont Health, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Enrollment Through 6 Months
Arm/Group | Autologous Muscle Derived Cells
Started | 23
Completed | 20
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: 6 Months Through 12 Months
Arm/Group | Autologous Muscle Derived Cells
Started | 20
Completed | 18
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Period: 12 Months Through End of Study
Arm/Group | Autologous Muscle Derived Cells
Started | 18
Completed | 17
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Of initial 23 subjects consented, 3 subjects withdrew from study prior to collection of initial data. Demographic data is not available for these 3 subjects.
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.45 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Study-related Adverse Events at 6 Months
Description: Safety of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by occurrences of study-related adverse events (AEs) reported by 6 months after enrollment. Number of reports of each adverse event is listed for events determined to be definitely or possibly related to study activities.
Time Frame: 6 months
Population: Participants may have reported more than one AE during this study period.
Measure: Number; unit: participants
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 20
participants
  Bruise | 2
  Pain | 1
  Scrotum discomfort | 1
  Scrotum swelling | 1
  Urinary tract infection | 1
  Vasovagal response | 1

2. Secondary Outcome: Number of Participants With Study-related Adverse Events Between 6 and 12 Months
Description: Long term safety of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by occurrences of study-related adverse events (AEs) reported between 6 and 12 months after enrollment. Number of reports of each adverse event is listed for events determined to be definitely or possibly related to study activities.
Time Frame: Between 6 and 12 months
Population: Subjects may have reported more than one adverse event during this study period
Measure: Number; unit: participants
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 20
participants
  Urine leakage | 1
  Bleeding at site of injection | 1

3. Secondary Outcome: Number of Participants With Improvement in Underactive Bladder Symptoms at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject completed GRA questionnaire. The GRA measures the subjects perceived level of change in underactive bladder symptoms at 12 months compared to before they were treated. The scale ranges from: Markedly worse, Moderately worse, Slightly worse, No change, Slightly improved, Moderately improved, to Markedly improved. Subjects select one response.
Time Frame: 12 months
Population: 17 subjects remaining in study at 12 months submitted data for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 17
Participants
  Markedly Improved | 0
  Moderately improved | 3
  Slightly improved | 9
  No change | 5
  Slightly worse | 0
  Moderately worse | 0
  Markedly worse | 0

4. Secondary Outcome: Number of Participants With Improvement in Underactive Bladder Symptoms at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject reported degree of change in urinary symptoms on the PGI-I at 12 months, compared to how their symptoms were before they began the study. Subjects select one response. The response scale ranges from: Very much better, Much better, A little bit better, No change, A little worse, Much worse, Very Much worse.
Time Frame: 12 months
Population: 17 subjects remaining in study at 12 months submitted data for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 17
Participants
  Very much better | 0
  Much better | 3
  A little bit better | 9
  No change | 5
  A little worse | 0
  Much worse | 0
  Very much worse | 0

5. Secondary Outcome: Change in Incontinence Questionnaire (ICIQ) Long Form Score From Baseline at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject reported urinary symptoms at 12 months from baseline. The ICIQ has a separate female (ICIQ-FLUTS Long form) and male (ICIQ-MLUTS long Form) set of questions to assess urinary symptoms in each sex. The total score range for ICIQ-FLUTS is 0-69. The total score range for ICIQ-MLUTS is 0-84. The sum of all the question scores equal a total score. Each question has a degree of bother scale associated with it. The degree of bother ranges from 0 (none at all) to 10 ( a great deal). Degree of bother scores are not incorporated in the overall score but indicate impact of the individual symptom. The difference taken in this analysis is the difference between the total score at 12 months minus the total score at baseline. If the difference is negative, it indicates improvement in the symptoms; 0 is no change; and a positive difference indicates a worsening of the symptoms.
Time Frame: 12 months
Population: 17 subjects remaining in the study at 12 months had data analyzed for this outcome: 3 female and 14 male.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 17
units on a scale
  Female (ICIQ-FLUTS) long form: number analyzed (Participants) | 3
  Female (ICIQ-FLUTS) long form | 0.6667 (5.1)
  Male (ICIQ-MLUTS) long form: number analyzed (Participants) | 14
  Male (ICIQ-MLUTS) long form | 1.071 (9.600)

6. Secondary Outcome: Change in Underactive Bladder Questionnaire (UABQ) Score From Baseline at 12 Months
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by subject reported changes to urinary symptoms at 12 months from baseline on the UABQ. The UABQ is a set of questions to assess urinary symptoms associated with underactive bladder. The total score ranges between 0 to 16. A lower score indicates a better outcome. A higher score indicates a worse outcome.
Time Frame: 12 months
Population: 17 subjects remaining at 12 months submitted data for analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 17
score on a scale | 5.7 (2.7)

7. Secondary Outcome: The Change in Number of Independent Voiding Occurrences Per Day on the 3-day Bladder Diary From Baseline at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject reported number of independent daytime voiding occurrences per day on the 3-day diary at 12 months compared to baseline. Positive numbers reflect a larger number of independent voids per day reported at baseline, and negative number represent a larger number of independent voids per day reported at 12 months.
Time Frame: 12 months
Population: 10 subjects had data available for both timepoints
Measure: Mean (Standard Deviation); unit: number of voids/day
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 10
number of voids/day | -0.665 (5.3)

8. Secondary Outcome: The Change in the Number of Voiding Occurrences Per Day Using a Catheter Recorded on the 3-day Bladder Diary From Baseline at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject reported number of daytime voiding occurrences per day using a catheter on the 3-day diary at 12 months compared to baseline. Positive numbers reflect a larger number of voiding occurrences per day reported at baseline, and negative numbers represent a larger number of voiding occurrences per day reported at 12 months.
Time Frame: 12 months
Population: 19 subjects had data reported for both timepoints
Measure: Mean (Standard Deviation); unit: number of voids/day
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 19
number of voids/day | -0.2094 (1.6)

9. Secondary Outcome: The Change in the Average Volume Voided Independently Per Day Measured in Milliliters Over the 3 Day Period Recorded on the 3-day Bladder Diary From Baseline at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject reported average volume voided independently per day over the 3 day period on the 3-day diary at 12 months compared to baseline. Volumes are measured in milliliters. Positive numbers reflect a larger volume voided per day at baseline, and negative numbers represent a larger volume voided per day at 12 months.
Time Frame: 12 months
Population: 10 subjects had data reported for both timepoints
Measure: Mean (Standard Deviation); unit: milliliters/day
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 10
milliliters/day | -156.66 (1100.0)

10. Secondary Outcome: The Change in the Average Volume in Milliliters Voided Per Day Using a Catheter Per Day Over the 3 Day Period Recorded on the 3-day Bladder Diary From Baseline at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject reported average volume voided using a catheter per day over the 3 day period on the 3-day diary at 12 months compared to baseline. Volumes are measured in milliliters. Positive numbers reflect a larger volume voided per day at baseline, and negative numbers represent a larger volume voided per day at 12 months.
Time Frame: 12 months
Population: 14 subjects had data for both timepoints
Measure: Mean (Standard Deviation); unit: milliliters/day
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 14
milliliters/day | -894.9 (2100)

11. Secondary Outcome: The Change in the Number of Bladder Leaks Over the 3 Day Period Recorded on the 3-day Bladder Diary From Baseline at 12 Months.
Description: The efficacy of Autologous Muscle Derived Cells in the treatment of underactive bladder as measured by changes to subject reported number of bladder leaks over the 3 day period on the 3-day diary at 12 months compared to baseline. Positive numbers reflect a larger number of leaks reported at baseline, and negative numbers represent a larger number of leaks reported at 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: bladder leaks per day
Arm/Group | Autologous Muscle Derived Cells
Number analyzed (Participants) | 20
bladder leaks per day | 0 (0)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Autologous Muscle Derived Cells
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Muscle Derived Cells (N=20)
Aortic stenosis (Cardiac disorders) | 1 (1)
Closed fracture of tibia (Musculoskeletal and connective tissue disorders) | 1 (1) — with fall
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Fracture of Humerus (Musculoskeletal and connective tissue disorders) | 1 (1) — with fall
Fracture of femoral neck (Musculoskeletal and connective tissue disorders) | 1 (1) — with fall
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Muscle Derived Cells (N=20)
Urinary tract infection (Renal and urinary disorders) | 10 (20)
Influenza (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bruise (Skin and subcutaneous tissue disorders) | 2 (2)
Fall (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02463448/Prot_SAP_000.pdf